CLINICAL TRIAL: NCT06301945
Title: Artificial Intelligence for Histopathological Classification and Recurrence Prediction of Thymic Epithelial Tumors
Brief Title: Artificial Intelligence Prediction Tool in Thymic Epithelial Tumors
Acronym: INTHYM
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maastro Clinic, The Netherlands (Other); Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Anna Salut Esteve Domínguez, PhD student, Erasmus Medical Center
Other Study IDs: Maastro Clinic; 72725524 (Other Grant/Funding Number: Hanarth Fonds)
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Thymic Epithelial Tumor; Thymic Carcinoma; Thymoma; Thymoma and Thymic Carcinoma
Keywords: Artificial Intelligence; Digital pathology
MeSH Terms: conditions — Thymic epithelial tumor; Thymoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with TET: Patients diagnosed with the following TET subtypes:
  * Thymoma Type A
  * Thymoma Type AB
  * Thymoma Type B1
  * Thymoma Type B2
  * Thymoma Type B3
  * Thymic Carcinoma
  Interventions: Diagnostic Test: Artificial Intelligence Diagnostics
- Recurrence: Patients with thymic epithelial tumors who have experienced recurrence.
  Interventions: Diagnostic Test: Recurrence Prediction Tool

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence Diagnostics — AI Diagnostics uses advanced algorithms for precise histological image analysis to help diagnose disease, including subtype.
  Other Names: AI Diagnostics, AI Classification
  Groups: Patients with TET
Diagnostic Test: Recurrence Prediction Tool — This AI tool evaluates thymic tumour data and other clinical data and calculates the risk of recurrence, with the aim of analysing whether there is an association with specific subtypes of thymic epithelial tumours and clinical data.
  Groups: Recurrence

SUMMARY:
Thymic epithelial tumors are rare neoplasms in the anterior mediastinum. The cornerstone of the treatment is surgical resection. Administration of postoperative radiotherapy is usually indicated in patients with more extensive local disease, incomplete resection and/or more aggressive subtypes, defined by the WHO histopathological classification.

In this classification thymoma types A, AB, B1, B2, B3, and thymic carcinoma are distinguished. Studies have shown large discordances between pathologists in subtyping these tumors. Moreover, the WHO classification alone does not accurately predict the risk of recurrence, as within subtypes patients have divergent prognoses.

The investigators will develop AI models using digital pathology and relevant clinical variables to improve the accuracy of histopathological classification of thymic epithelial tumors, and to better predict the risk of recurrence.

In this multicentric and international project three existing databases will be used from Rotterdam, Maastricht and Lyon. For all models one database will be used to build AI models, and the other two for external validation.

The ultimate goal of this project is to develop AI models that support the pathologist in correctly subtyping thymic epithelial tumors, in order to prevent patients from under- or overtreatment with adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Participants with specific diagnoses are eligible for inclusion in the study. The eligible diagnoses include various subtypes of thymoma and thymic carcinoma, specifically:

* Thymoma A
* Thymoma AB
* Thymoma B1
* Thymoma B2
* Thymoma B3
* Thymic Carcinoma

Inclusion is based on a consensus diagnosis with a level of agreement less than 70%. This criterion is applied during the training phase of the model.

Recurrence Criteria:

Participants with a documented recurrence outcome within a 5-year period are considered eligible for this aspect of the study. This criterion is primarily applied during the validation phase.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study Population:
  This study focuses on individuals diagnosed with thymic epithelial tumors. The study includes patients from three datasets: Erasmus MC (710 patients), Maastro (137 patients), and University Hospital Lyon (181 patients).
  Additional Information:
  * Erasmus MC (710 patients): Includes age, gender, and diagnosis information; each patient may have multiple whole slide images.
  * Maastro (137 patients): Each patient may have multiple whole slide images.
  * University Hospital Lyon (181 patients): Each patient may have multiple whole slide images.
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
WP1 - Databases/Data Pre-processing | M1-M18
  The EMC-dataset includes 179 TET-patients classified by experienced TET-pathologists. Cases with good agreement between pathologists will be used for training AI-models. Evaluation includes digitized pathology slides assessed by an international expert-panel. The MUMC-database (137 patients) and CHUL-database (181 patients) provide additional data, including clinical variables. Relevant factors include age, gender, tumor volume, stage, completeness of resection, autoimmune disorders, and treatment details.

SECONDARY OUTCOMES:
WP2 - Deep Learning-Model for TET Classification and Recurrence Prediction | M6-M32
  This outcome aims to create an AI-framework with two principal goals. First, investigate TET-subtypes using four different models emphasizing cell type, morphological structures, and a combination. Second, classify patients based on recurrence outcome within 5 years. An ablation study will be conducted with state-of-the-art deep learning classifiers (ResNet, Inception).

OTHER OUTCOMES:
WP3: Clinical Evaluation | M6-M36
  AI-models 1-3 will be built and validated on the EMC-database, while AI-model 4 will be built on the MUMC+-database and validated on both. Model performance will be assessed using sensitivity, specificity, negative/positive predictive value. Decision analysis curves will quantify the clinical benefit, identifying patient groups with the largest utility.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf JL, van Nederveen F, Blaauwgeers H, Marx A, Nicholson AG, Roden AC, Strobel P, Timens W, Weissferdt A, von der Thusen J, den Bakker MA. Interobserver variation in the classification of thymic lesions including biopsies and resection specimens in an international digital microscopy panel. Histopathology. 2020 Nov;77(5):734-741. doi: 10.1111/his.14167. Epub 2020 Sep 24. PMID 32506527
- [Background] Molina TJ, Bluthgen MV, Chalabreysse L, de Montpreville VT, de Muret A, Dubois R, Hofman V, Lantuejoul S, le Naoures C, Mansuet-Lupo A, Parrens M, Piton N, Rouquette I, Secq V, Girard N, Marx A, Besse B. Impact of expert pathologic review of thymic epithelial tumours on diagnosis and management in a real-life setting: A RYTHMIC study. Eur J Cancer. 2021 Jan;143:158-167. doi: 10.1016/j.ejca.2020.11.011. Epub 2020 Dec 11. PMID 33316754